CLINICAL TRIAL: NCT00259909
Title: A Prospective Observational Study for the Psychometric Validation of a Patient-reported Questionnaire in Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD)
Brief Title: Observational Study Of An Electronic Questionnaire In Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: OPL104226
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Infections, Bacterial
Keywords: Patient reported outcomes; COPD; acute exacerbation of chronic obstructive pulmonary disease (AECOPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with COPD: Subject has a confirmed clinical diagnosis of COPD, with or without chronic bronchitis.
  Interventions: Other: GSK questionnaire; Other: St. George's Respiratory Questionnaire; Other: Acute Short Form 12 version 2; Other: Global Efficacy questionnaire

INTERVENTIONS:
Other: GSK questionnaire — GSK questionnaire will demonstrate the validity, reliability and responsiveness as a tool for measuring subject-reported outcomes during an acute exacerbation of chronic obstructive pulmonary disease.
Other: St. George's Respiratory Questionnaire — The SGRQ is a 50-item questionnaire with 76 weighted responses. It provides a Total score and three component scores: Symptoms (distress caused by respiratory symptoms), Activity (physical activities that cause or are limited by breathlessness), and Impacts (social and psychological effects of the disease). The Total score and each of the SGRQ sub-scores are scored from 0 to 100 where 0 indicates best and 100 indicates worst health.
Other: Acute Short Form 12 version 2 — The Acute SF-12v2 is a multipurpose short-form questionnaire with only 12 questions with two summary scores, the SF-12 Physical Component Summary (PCS-12) and the SF-12 Mental Component Summary (MCS-12). The scoring range for the PCS-12 and MCS-12 is 0 to 100, with a lower score indicating a poorer level of health
Other: Global Efficacy questionnaire — Global Efficacy questionnaire will be administered in an electronic form to validate test-retest reliability, responsiveness and minimum important difference (MID)

SUMMARY:
The aim of the study is to develop a new patient-reported outcome (PRO) questionnaire measuring the impact of an acute exacerbation on daily lives of patients with chronic obstructive pulmonary disease (COPD). This questionnaire will aim to detect an acute exacerbation and resolution of exacerbation from the patient's perspective. At a later stage of development, this questionnaire will be able to measure the effect of anti bacterials in the treatment of acute exacerbations of COPD (AECOPD). This study will evaluate the factor structure, validity, reliability, and responsiveness of the GSK questionnaire in subjects who experience acute exacerbations of their COPD.

ELIGIBILITY:
Inclusion Criteria:

* 15 pack-year smoking history.
* Confirmed diagnosis of COPD.
* Have two documented episodes of acute exacerbation in past 12 months.

Exclusion Criteria:

* Clinical diagnosis of asthma.
* Subjects not literate in the language of the questionnaire (e.g. US English).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject has a confirmed clinical diagnosis of COPD, with or without chronic bronchitis were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2005-11-02 (Actual); Primary Completion 2006-11-07 (Actual); Study Completion 2006-11-07 (Actual)

PRIMARY OUTCOMES:
St. George's Respiratory Questionnaire (SGRQ) Scores at Baseline | Day 1
  The SGRQ is a 50-item questionnaire with 76 weighted responses. It provides a Total score and three component scores: Symptoms (distress caused by respiratory symptoms), Activity (physical activities that cause or are limited by breathlessness), and Impacts (social and psychological effects of the disease). The Total score and each of the SGRQ sub-scores are scored from 0 to 100 where 0 indicates best and 100 indicates worst health. An increase in score indicates worsening health. A change in the Total score of 4 units is consistent with a clinically significant change in the subject
SGRQ Scores at exacerbation | Up to Day 14
  The SGRQ is a 50-item questionnaire with 76 weighted responses. It provides a Total score and three component scores: Symptoms (distress caused by respiratory symptoms), Activity (physical activities that cause or are limited by breathlessness), and Impacts (social and psychological effects of the disease). The Total score and each of the SGRQ sub-scores are scored from 0 to 100 where 0 indicates best and 100 indicates worst health. An increase in score indicates worsening health. A change in the Total score of 4 units is consistent with a clinically significant change in the subject
SGRQ Scores post-exacerbation | Up to Day 14
  The SGRQ is a 50-item questionnaire with 76 weighted responses. It provides a Total score and three component scores: Symptoms (distress caused by respiratory symptoms), Activity (physical activities that cause or are limited by breathlessness), and Impacts (social and psychological effects of the disease). The Total score and each of the SGRQ sub-scores are scored from 0 to 100 where 0 indicates best and 100 indicates worst health. An increase in score indicates worsening health. A change in the Total score of 4 units is consistent with a clinically significant change in the subject
Acute Short Form 12 version 2 (Acute SF-12v2) scores at Baseline | Day 1
  The Acute SF-12v2 is a multipurpose short-form questionnaire with only 12 questions with two summary scores, the SF-12 Physical Component Summary (PCS-12) and the SF-12 Mental Component Summary (MCS-12). The scoring range for the PCS-12 and MCS-12 is 0 to 100, with a lower score indicating a poorer level of health. It has been translated and validated in most major languages. The Acute SF-12v2 is self-administered by patients, and completed on average in 2 minutes or less.
Acute SF-12v2 scores at exacerbation | Up to Day 14
  The Acute SF-12v2 is a multipurpose short-form questionnaire with only 12 questions with two summary scores, the SF-12 Physical Component Summary (PCS-12) and the SF-12 Mental Component Summary (MCS-12). The scoring range for the PCS-12 and MCS-12 is 0 to 100, with a lower score indicating a poorer level of health. It has been translated and validated in most major languages. The Acute SF-12v2 is self-administered by patients, and completed on average in 2 minutes or less.
Acute SF-12v2 scores post-exacerbation | Up to Day 14
  The Acute SF-12v2 is a multipurpose short-form questionnaire with only 12 questions with two summary scores, the SF-12 Physical Component Summary (PCS-12) and the SF-12 Mental Component Summary (MCS-12). The scoring range for the PCS-12 and MCS-12 is 0 to 100, with a lower score indicating a poorer level of health. It has been translated and validated in most major languages. The Acute SF-12v2 is self-administered by patients, and completed on average in 2 minutes or less.
Global Efficacy questionnaire scores at Baseline | Day 1
  Global Efficacy questionnaire will be administered in an electronic form to validate test-retest reliability, responsiveness and minimum important difference (MID)
Global Efficacy questionnaire scores at exacerbation | Up to Day 14
  Global Efficacy questionnaire will be administered in an electronic form to validate test-retest reliability, responsiveness and minimum important difference (MID)
Global Efficacy questionnaire scores post-exacerbation | Up to Day 14
  Global Efficacy questionnaire will be administered in an electronic form to validate test-retest reliability, responsiveness and minimum important difference (MID)
Physician reported measures at Baseline | Day 1
Physician reported measures at exacerbation | Up to Day 14
Physician reported measures post-exacerbation | Up to Day 14

SECONDARY OUTCOMES:
Change from Baseline in SGRQ-C Total and Subscales Scores | Up to Day 14
Percentage change in SGRQ-C scores | Up to Day 14
Change from Baseline in Acute SF-12v2 Total and Subscales Scores | Up to Day 14
Percentage change in Acute SF-12v2 scores | Up to Day 14
Change from Baseline in Global Efficacy Questionnaire Total and Subscales Scores | Up to Day 14
Percentage change in Global Efficacy Questionnaire scores | Up to Day 14
Change from Baseline in GSK questionnaire Total and Subscales Scores | Up to Day 14
Percentage change in GSK questionnaire scores | Up to Day 14
Time to resolution of each domain score | Up to Day 35
Time to resolution of total domain score | Up to Day 35

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (105):
- United States (72):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Hueytown, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Hines, Illinois
  - GSK Investigational Site, North Chicago, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Newburgh, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Dubuque, Iowa
  - GSK Investigational Site, Waterloo, Iowa
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, DeWitt, Michigan
  - GSK Investigational Site, Plainwell, Michigan
  - GSK Investigational Site, Richland, Michigan
  - GSK Investigational Site, Saint Joseph, Michigan
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Kirkwood, Missouri
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, East Brunswick, New Jersey
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Kingston, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Audubon, Pennsylvania
  - GSK Investigational Site, King of Prussia, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Plymouth Meeting, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Morristown, Tennessee
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Germany (19):
  - GSK Investigational Site, Schwetzingen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Bad Woerrishofen, Bavaria
  - GSK Investigational Site, Kötzting, Bavaria
  - GSK Investigational Site, Landsberg am Lech, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Euskirchen, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Lüdenscheid, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Wahlstedt, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (14):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Caserta, Campania
  - GSK Investigational Site, Eboli (SA), Campania
  - GSK Investigational Site, Salerno, Campania
  - GSK Investigational Site, Telese Terme (BN), Campania
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Rozzano (MI), Lombardy
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, San Martino in Tregnano (Spoleto, PG), Umbria
  - GSK Investigational Site, San Sisto (PG), Umbria
  - GSK Investigational Site, Spoleto (PG), Umbria
  - GSK Investigational Site, Cittadella (PD), Veneto